CLINICAL TRIAL: NCT03693820
Title: The Effect of Gallbladder Bed Infiltration on Analgesia in Laparoscopic Cholecystectomy
Brief Title: Gall Bladder Bed Infiltration Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alaa Mazy Mazy (Other)
Responsible Party: Sponsor-Investigator, Alaa Mazy Mazy, associate prosseor, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MS.18.09.277
Record Dates: First submitted 2018-10-01; First posted 2018-10-03 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2018-10

CONDITIONS: Pain, Acute
Keywords: cholecystectomy;; analgesia;; gallbladder;; infiltration;; visceral pain
MeSH Terms: conditions — Acute Pain; Agnosia; Visceral Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: the infiltration cocktail of local anesthetic will be replaced by saline in the same volume.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the infiltration group (Active Comparator): a cocktail of 5 mg/Kg lidocaine normal saline in a volume of 3 ml/Kg 5 mcg/ml adrenaline. We will administrate 5 ml lidocaine at each port site before incision, then immediately after the creation of the pneumoperitoneum, the surgeon will spray 50-75 ml of the total solution on the upper surface of the liver under the right sub-diaphragmatic space and another 50-75ml over the parietal peritoneum. The Trendelenburg position will be maintained for 2 minutes. Then 50 ml will be infiltrated in the bladder bed and pedicle after clamping of the cystic duct and artery. Infiltration will be through a laparoscopic suction needle, diameter 0.9 /330 mm (Zhejiang, China).
  Interventions: Drug: the infiltration group
- the control group (Placebo Comparator): the same technique but the 50 ml for gallbladder infiltration will be replaced by saline.
  Interventions: Drug: the control group

INTERVENTIONS:
Drug: the infiltration group — * 15-20 ml periportal,
  * 50 ml in gallbladder bed,
  * The rest (about 150 ml in 70 Kg patient) will be intraperitoneal
  Arms: the infiltration group
Drug: the control group — the 50 ml prepared for gallbladder bed infiltration will be replaced by saline.
  Arms: the control group

SUMMARY:
Early postoperative pain is a common complaint after elective laparoscopic cholecystectomy. Persistent acute postoperative pain is the dominating complaint and the primary reason for a prolonged stay after this procedure. This pain can be superficial incisional wound pain (somatic), deep visceral pain and/or post-laparoscopy shoulder pain (referred somatic), all of which may require systemic analgesia. Hypothesis: Laparoscopic pain can be superficial incisional wound pain (somatic pain), deep visceral pain and/or post-laparoscopy shoulder pain (referred somatic pain), so the block must be periportal for incisional wound pain, intraperitoneal to decrease pain caused by pneumoperitoneum, and of the bladder bed to decrease the deep visceral pain. This combination can give the maximum analgesia after laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Bladder bed irrigation with Bupivacaine was an effective method for reducing pain during the first postoperative hours after laparoscopic cholecystectomy. The intraperitoneal administration of lidocaine solution (total dose, 3.5 mg/kg) will be done as follows: immediately after creation of the pneumoperitoneum, the surgeon will spray 50-75 ml of the total solution on the upper surface of the liver under the right sub-diaphragmatic space, and another 50-75ml of the total solution under the left sub-diaphragmatic space. In order to allow the sprayed solution to diffuse under the diaphragmatic space, the Trendelenburg position will be maintained for 2 minutes.

In the infiltration group will be administrating 5 ml lidocaine at each port site before incision, then the surgeon will spray 50-75 ml of the total solution on the upper surface of the liver under the right sub-diaphragmatic space, and another 50-75ml of the total solution under the left sub-diaphragmatic space then 50 ml will be infiltrated in the bladder bed after clamping of the cystic duct and cystic artery. CO2 will be humidified and wormed.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo elective laparoscopic cholecystectomy.
* American Society of Anesthesiologists physical status (ASA) I or II.

Exclusion Criteria:

1. Patient in receipt of analgesics or sedatives 24 h before scheduled surgery.
2. Patient with spillage or cholelithiasis with known common bile duct pathology.
3. Body Mass Index > 40 Kg/m2.
4. Patient underlying severe systemic disease.
5. Patient with a history of abdominal surgery, a chronic pain disorder other than gallbladder disease or allergy to lidocaine.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-07-11 (Actual)

PRIMARY OUTCOMES:
The total postoperative analgesic consumption | postoperative, for 24 hours
  ketorolac and morphine in mg .

SECONDARY OUTCOMES:
The time to the first request of analgesia | postoperative, for 24 hours
  hours
The intraoperative fentanyl requirements. | intraoperative
  microgram
postoperative pain score: VAS | postoperative at 0, 2, 4, 8, 12, 16 and 24 hours
  visual analog score from 0-10, zero is no pain, 10 is the most imaginable pain,
heart rate | basal and intraoperatively every 30 minutes, then at 0, 2, 4, 8, 12, 16 and 24 hours post-operatively.
  beat/ minute
mean blood pressure | basal and intraoperatively every 30 minutes, then at 0, 2, 4, 8, 12, 16 and 24 hours post-operatively.
  mmHg
incidence of vomiting | postoperatively, during the first 24 hours
  number
the sleep quality | postoperatively, after the first night.
  through a score 0-2, where 0= good quite sleep, 1= fair sleep, 2= bad quality of sleep.
Patient satisfaction regards analgesia: | postoperative after 24 hour.
  using visual analog score from 0-10. zero = no satisfaction, 12= maximum satisfaction.
Surgeon satisfaction regards the technique: | postoperative within 1 hour.
  using visual analog score from 0-10. zero = no satisfaction, 10= maximum satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: alaa mazy, MD, Study Director — faculty of medicine, Mansoura
Locations (1):
- Gastro-enterolgy surgical center, Mansoura University, Al Mansurah, Al-Dakahleia, Egypt